CLINICAL TRIAL: NCT05375032
Title: Acute Effects of Cycling Dual-task on Cognitive and Physical Function in Parkinson´s Disease: a Cross-sectional Study.
Brief Title: Acute Effects of Cycling Dual-task in Parkinson´s Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Iris Machado de Oliveira, Principal Investigator, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205-2022-2
Record Dates: First submitted 2022-05-02; First posted 2022-05-16 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cycling combined with cognitive tasks (Experimental)
  Interventions: Other: Cycling combined with cognitive tasks
- Cycling (Active Comparator)
  Interventions: Other: Cycling

INTERVENTIONS:
Other: Cycling combined with cognitive tasks — A 30-minute session of Forced Cycling aerobic exercise performed with lower limbs and free active cycling performed with upper limbs combined with cognitive stimuli. An intelligent cycle ergometer (Motomed Viva 2 Parkinson) will be used, at a reserve heart rate of 55-70% (Borg scale 12-14) during the active part. The forced cycling program will consist of a 6-minute passive warm-up part (40-60 RPM), a 20-minute active part (90 RPM), and a 4-minute passive cool down (40 RPM). The cognitive task will be a PowerPoint presentation structured in a way that is consistent with the phases of the cycling program. The passive phases (6 minutes of warm-up and 4 minutes of passive cycling back to cool down), images of the nearby environment will be played. For the active phase (20 minutes of assisted active cycling) the PowerPoint presentation will be structured with tasks related to: orientation, memory, calculation, language, similarities.
  Other Names: Cycling dual task
  Arms: Cycling combined with cognitive tasks
Other: Cycling — A 30-minute session of Forced Cycling aerobic exercise performed with lower limbs and free active cycling performed with upper limbs combined with cognitive stimuli. An intelligent cycle ergometer (Motomed Viva 2 Parkinson) will be used, at a reserve heart rate of 55-70% (Borg scale 12-14) during the active part. The forced cycling program will consist of a 6-minute passive warm-up part (40-60 RPM), a 20-minute active part (90 RPM), and a 4-minute passive cool down (40 RPM).
  Arms: Cycling

SUMMARY:
Taking into account the process of functional and cognitive evolution that patients with Parkinson's disease experience throughout the pathology, the objective of this study is to evaluate the acute effects of aerobic exercise in forced cycling performed with lower limbs and freecycling of upper limbs combined with cognitive stimuli on attention, exploration skills, and short-term motor skills in people with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease
* Present stage between I and III on the Hoenh and Yarh scale
* Being able to move autonomously

Exclusion Criteria:

* Moderate-severe cognitive impairment (Mini-mental test > 24)
* Comorbidity that discourages the practice of physical exercise and that allows performing all scheduled assessments
* Severe visual alterations that prevent the development of the session

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline Symbol Digit Modalities Test at 30 minutes | Pre and up to 30 minutes.
  Detection of cognitive dysfuntions.
Mini-Mental State Examination (MMSE) | Pre
  To detect and estimate cognitive decline and dementia.

SECONDARY OUTCOMES:
Borg Rated Perceived Exertion Scale | Up to 30 minutes.
  Perceived exertion. These include a rating of 6 perceiving "no exertion at all" to 20 perceiving a "maximal exertion" of effort.
Change from baseline Heart Rate at 30 minutes | Pre and up to 30 minutes
  Heart rate

OTHER OUTCOMES:
Active Distance (m) | During the unique session
  Cycling active distance in meters.
Passive Distance (m) | During the unique session
  Cycling assisted distance in meters.
Total Work (W) | During the unique session
  Cycling total work developed in Watts
Active Speed (rpm) | During the unique session
  Average cycling active speed in rotation per minute
Passive Speed (rpm) | During the unique session
  Average cycling assisted speed in rotation per minute
Symmetry (%) | During the unique session
  Percentage of the active work developed by each lower limb, right and left.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vigo, Pontevedra, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No